CLINICAL TRIAL: NCT06778369
Title: Triangular Exclusion Technique in Isolated Posterior Mitral Valve Leaflet Prolapse for Mitral Valve Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sameh Elsayed Saeed Elsayed, lecturer, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB # 11120-20-9-2023
Record Dates: First submitted 2024-12-27; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Mitral Valve Posterior Leaflet Prolapse
Keywords: Mitral valve repair;Triangular Exclusion Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- traingular exclusion technique (Experimental): Triangular exclusion technique in isolated posterior mitral valve leaflet prolapse for mitral valve repair
  Interventions: Procedure: traingular exclusion technique in mitral valve repair

INTERVENTIONS:
Procedure: traingular exclusion technique in mitral valve repair — The prolapsed part of the posterior leaflet is inverted and excluded, not resected toward the left ventricle, and the margins of the prolapsed part are sutured to each other's using proline 5/0, extending from the posterior leaflet edge to the posterior annulus. Then the posterior annulus is reinforced with an annuloplasty band using a treated strip of pericardium. The determination of suitable ring size is subsequently predicated upon the assessment of inter-commissural distance surface area and the anterior leaflet, utilizing sizers that are correlated with typical mitral geometry.

SUMMARY:
The goal of this clinical trial is to learn if surgical method done to repair one of the heart valve called mitral valve disease during open heart surgery

The main questions aims to answer is:

Does this method is safe and effective for long time and can be used in special cases of mitral valve surgery ? participants come to clinic to be checked clinically and radiologcally every month by the surgeon till 12 month

DETAILED DESCRIPTION:
the surgical method isThe prolapsed part of the posterior leaflet of the mitral valve is inverted and excluded, toward the left ventricle but not cutted echocardiography done before participants leave hospital after sugery, after 6 month and after 12 months to confirm that this method of repair is safe and effective for participants life long

ELIGIBILITY:
Inclusion Criteria:

* varying degrees of degenerative MV regurgitation, ranging from moderate to severe or severe caused by isolated prolapse of the posterior MV leaflet
* concomitant tricuspid annuloplasty

Exclusion Criteria:

* with Mitral Valve stenosis or any other manifestation of mitral regurgitation pathology.
* individuals requiring surgical intervention for the aortic or pulmonary valves

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
degree of postoperative mitral valve regurgitation following Triangular Exclusion Technique | about 13 months From enrolment to the end of surgical procedure about one month follow up Echo done after 6 and 12 months so total time frame about 13 months duration
  Suggested Quality Metrics for Interventions for Mitral Regurgitation
  1. Procedural success Absence of moderate or worse residual mitral regurgitation (on TTE within 30 days) Absence of stroke or mortality
  2. Procedural effectiveness (1 year) Alive Freedom from moderate or worse mitral regurgitation Freedom from cardiovascular reintervention Freedom from NYHA functional class III-IV symptoms
  3. Durability (5 years or later) Freedom from moderate or worse mitral regurgitation Freedom from mitral valve reintervention But our study limited to only 1 year follow up due to our academic authorities that will be added as one of the strong limitations of our study but we will mention at conclusion and recommendations to extend the sample size and follow up period of the operated patients till 5 years in the following studies that interested by the same topic

CONTACTS AND LOCATIONS:
Overall Officials: sameh saeed, lecturer, Principal Investigator — cardiothoracic surgery department-faculty of medecine-Zagazig univeristy-Egypt
Locations (1):
- cardiothorathic surgery department -faculty of medecine-zagazig univeristy-Egypt, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No